CLINICAL TRIAL: NCT06925295
Title: Image-Based Functionally Adapted Radiation Therapy for Lung Cancer
Brief Title: Using Xe MRI to Guide Radiation Therapy for Lung Cancer
Acronym: (XeRTLC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sean Fain (Other)
Responsible Party: Sponsor-Investigator, Sean Fain, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202408283
Record Dates: First submitted 2025-03-28; First posted 2025-04-13 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Imaging Techniques
Keywords: Lung cancer; Xenon; Imaging
MeSH Terms: conditions — Lung Neoplasms | interventions — Respiratory Function Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Technical Development Arm (Experimental): Lung cancer patients who will undergo standard-of-care stereotactic body radiation therapy (SBRT).
  Interventions: Drug: Xenon MRI; Diagnostic Test: Pulmonary Function Testing; Other: Quality of Life Questionnaire; Other: Medical Research Council Dyspnea score; Other: St. George's Respiratory Questionnaire; Diagnostic Test: Blood Biomarkers
- Implementation Arm (Experimental): Lung cancer patients who will undergo SBRT plans that were functionally adapted to avoid highly functioning lung based on Xe MRI.
  Interventions: Drug: Xenon MRI; Diagnostic Test: Pulmonary Function Testing; Other: Quality of Life Questionnaire; Other: Medical Research Council Dyspnea score; Other: St. George's Respiratory Questionnaire; Diagnostic Test: Blood Biomarkers

INTERVENTIONS:
Drug: Xenon MRI — MRI with Xenon used for contrast
Diagnostic Test: Pulmonary Function Testing — Pulmonary function testing will include spirometry, lung volumes, DLCO and oscillometry
Other: Quality of Life Questionnaire — European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30+QLQ-LC29)
Other: Medical Research Council Dyspnea score — modified Medical Research Council Dyspnea score (mMRC Dyspnea)
Other: St. George's Respiratory Questionnaire — St. George's Respiratory Questionnaire (SGRQ)
Diagnostic Test: Blood Biomarkers — blood biomarkers of inflammation and injury (e.g. Angiopoetin-2, Interleukin-6, myofibroblast activity, BPD4)

SUMMARY:
The purpose of this research study is to explore using MRI scans with xenon to better image lung function, how lung function changes after radiation therapy, and to guide radiation therapy away from parts of the lung that have good function. This project is foundational to performing additional studies to establish if novel MRI imaging can serve as a guidance tool for lung cancer radiation treatment.

DETAILED DESCRIPTION:
Despite the recent implementation of daily adaptation of image-guided radiation treatment using highly precise beam delivery technologies, significant acute and chronic lung toxicity is still reported in approximately 20% of lung cancer patients undergoing radiation therapy. Furthermore, subclinical loss of lung function is a concern for long term outcomes and quality of life. The purpose of this pilot study is to develop, implement and evaluate the efficacy of a new radiation therapy (RT) treatment planning paradigm that incorporates regional pulmonary functional imaging information to reduce radiation dose to healthy lung tissues.

The central hypothesis is that functional lung magnetic resonance imaging (MRI) using hyperpolarized xenon (Xe) will provide the means to visualize and quantify acute ventilation and gas exchange alterations during a standard course of RT treatment, and that modifying radiation treatment plans based on the combination of functional and anatomical MRI will result in improved outcomes for lung cancer patients in the short and long term. The rationale for the proposed research is that the implementation of functional imaging context into RT treatment planning is currently inhibited by a lack of access to routine MRI-guidance and a robust workflow to practically incorporate functional information into clinical treatment planning.

The study has the following Specific Aims: 1) Develop automated software tools to integrate functional Xe MRI into RT treatment planning software and establish a comprehensive clinical workflow to reduce radiation dose in highly-functioning regions of the lung, 2) Monitor the acute and chronic effects of RT on lung ventilation and gas exchange using Xe MRI and identify early functional imaging biomarkers of radiation induced lung injury, and 3) Compare outcomes and the post-treatment trajectory of pulmonary functional measurements between functional MRI-guided and standard RT cohorts to assess the potential efficacy of Xe MRI guided adaptive RT. The overall scientific objective is to develop a comprehensive workflow that enables functional lung sparing and monitoring of acute and chronic (6 months post RT) pulmonary functional injury in lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the trial

1. Aged 18-80 years
2. Willing and able to provide informed consent and adhere to visit/protocol schedules (Consent must be given before any study procedures are performed.)
3. Clinical diagnosis of lung cancer made by a board-certified oncologist with intent to treat with stereotactic body radiation therapy. We will not exclude individuals based on cancer type or severity of disease with the exception of the below criteria

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the trial:

1. Subject is less than 18 years old or incarcerated
2. MRI is contraindicated based on responses to MRI screening questionnaire
3. Subject is pregnant or lactating
4. Resting oxygen saturation <90% on supplemental oxygen
5. Respiratory illness of bacterial or viral etiology within 30 days of planned treatment
6. Subject has history of any known ventricular cardiac arrhythmia
7. Subject has history of cardiac arrest within the last year
8. Subject has prior history of cancer treatment with radiation therapy to the lung
9. Subject has concurrent cancer treatment with agents associated with increased risk of radiation pneumonitis (e.g. immunotherapy, chemotherapy)
10. Subject does not fit into 129Xe vest coil used for MRI
11. Subject cannot hold his/her breath for 15 seconds
12. Subject deemed unlikely to be able to comply with instructions during imaging
13. Medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of PFT evidence of radiation pneumonitis and lung function change on spirometry | Baseline Visit, periprocedural, 1 month follow up visit, and 6 month follow up visit..
  is the incidence of PFT evidence of radiation pneumonitis and lung function change. Change in spirometry will be reported as the mean±SD of these measurements for each treatment study visit, and the mean difference of these measurements from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Fain, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided